CLINICAL TRIAL: NCT01058733
Title: Seoul St. Mary's Hospital College of Medicine The Catholic University of Korea, Seoul, Korea
Brief Title: Semi-automatic Response System(SARS)in Type 2 Diabetes
Acronym: SARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Kun-Ho Yoon, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARS-Project
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus
Keywords: semi-automatic response system (SARS); Diabetes Mellitus; Internet; ubiquitous health care system
MeSH Terms: conditions — Diabetes Mellitus | interventions — Patient Portals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Internet (Other): New clinical decision-supporting system for glucose monitoring, SARS, which could identify glucose data recorded by patients and make some optimal decisions.The SARS engine assigned subjects to one of three levels according to the glucose control status and glucose control method.
  Interventions: Other: Internet

INTERVENTIONS:
Other: Internet — new clinical decision-supporting system for glucose monitoring, SARS, which could identify glucose data recorded by patients and make some optimal decisions.The SARS engine assigned subjects to one of three levels according to the glucose control status and glucose control method.
  Other Names: clinical decision-supporting system

SUMMARY:
Background

* Various kinds of interactive online communication systems have been introduced for long-term diabetes management, and their importance in managing patients is increasing. The investigators investigated the amount of physician time needed to maintain such a system, and the investigators developed software to maximise the cost effectiveness.

Methods

* The investigators conducted a prospective, randomised, controlled trial to investigate the efficacy and safety of a semi-automatic response system (SARS) for online glucose monitoring over a 24-week period of patients with type 2 diabetes. In the SARS group, the "SARS" software filtered the recorded self-monitoring of blood glucose data automatically to reduce the physicians' time, and the physicians managed patients regularly but only manually in the control (manual) group. The investigators measured the time spent by the physicians for online management and compared the HbA1c levels at enrolment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* men or women aged 20-70 years with type 2 diabetes
* lasting more than one year who had used the online communication system for diabetes management at the web site https://www.bi odang.com for more than six months
* baseline HbA1c level was 6-10%
* Patients who able and willing to complete glucose-monitoring diaries on a web chart as instructed.

Exclusion Criteria:

* patients who required intensive insulin therapy (multiple insulin injections or insulin pump therapy) or who were unwilling to use self-monitoring of blood glucose (SMBG)
* acute metabolic complications of diabetes (e.g., diabetic ketoacidosis, hyperosmolar non-ketotic hyperglycaemia, lactic acidosis)
* serum creatinine concentration >2.0 mg/dl at screening
* active liver disease or ALT or AST activities >2.5 times the upper limit of normal
* acute illness, chronic infection, heart failure of NYHA Class III or IV
* recent myocardial infarction or stroke during the past six months
* pregnancy or GDM, or any other factor likely to limit protocol compliance or reporting of adverse events

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
physicians' labour time and frequency of contact with the online communication system required for reviewing the patients' information and sending recommendations | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, Principal Investigator — Seoul St. Mary's Hospital, Seoul, Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Kwon HS, Cho JH, Kim HS, Song BR, Ko SH, Lee JM, Kim SR, Chang SA, Kim HS, Cha BY, Lee KW, Son HY, Lee JH, Lee WC, Yoon KH. Establishment of blood glucose monitoring system using the internet. Diabetes Care. 2004 Feb;27(2):478-83. doi: 10.2337/diacare.27.2.478. PMID 14747232
- [Background] Yoon KH, Lee JH, Kim JW, Cho JH, Choi YH, Ko SH, Zimmet P, Son HY. Epidemic obesity and type 2 diabetes in Asia. Lancet. 2006 Nov 11;368(9548):1681-8. doi: 10.1016/S0140-6736(06)69703-1. PMID 17098087
- [Background] Kwon HS, Cho JH, Kim HS, Lee JH, Song BR, Oh JA, Han JH, Kim HS, Cha BY, Lee KW, Son HY, Kang SK, Lee WC, Yoon KH. Development of web-based diabetic patient management system using short message service (SMS). Diabetes Res Clin Pract. 2004 Dec;66 Suppl 1:S133-7. doi: 10.1016/j.diabres.2003.10.028. PMID 15563964
- [Background] Cho JH, Chang SA, Kwon HS, Choi YH, Ko SH, Moon SD, Yoo SJ, Song KH, Son HS, Kim HS, Lee WC, Cha BY, Son HY, Yoon KH. Long-term effect of the Internet-based glucose monitoring system on HbA1c reduction and glucose stability: a 30-month follow-up study for diabetes management with a ubiquitous medical care system. Diabetes Care. 2006 Dec;29(12):2625-31. doi: 10.2337/dc05-2371. PMID 17130195
- [Background] Cho JH, Lee HC, Lim DJ, Kwon HS, Yoon KH. Mobile communication using a mobile phone with a glucometer for glucose control in Type 2 patients with diabetes: as effective as an Internet-based glucose monitoring system. J Telemed Telecare. 2009;15(2):77-82. doi: 10.1258/jtt.2008.080412. PMID 19246607